CLINICAL TRIAL: NCT02272257
Title: Direct Access Physical Therapy Compared With Physician Portal of Entry for Temple University Employees With Recent Onset Musculoskeletal Conditions: A Randomized Controlled Trial.
Brief Title: Temple University Employees With Musculoskeletal Conditions Receive Physical Therapy to Treat Limitations Early
Acronym: TEMPLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 22290
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-04

CONDITIONS: Musculoskeletal Diseases
Keywords: Musculoskeletal Pain; Physical Therapists; Drug Prescriptions; Humans; Physical Therapy Modalities; Referral and Consultation; Workers' Compensation; United States; Primary Care; Health Services Research; Triage; Acute; Cost; Occupational Health
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain | interventions — Practice Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Direct Access Physical Therapy (Experimental): All care will be administered by one or more physical therapists employed by Temple University. This arm will be early, direct access, physical therapy (immediately evaluation following contacting the front desk administrator or reporting a work injury). Intervention will include interventions matched to their stratified risk category incorporating biopsychosocially oriented education, therapeutic exercise, and manual therapy tailored to the patient's needs.
  Interventions: Behavioral: Early Direct Access Physical Therapy
- Physician management (Active Comparator): All usual care by physician will be administered by one or more employee health physicians employed by Temple University. Recommendations may or may not include referral to physical therapy.
  Interventions: Behavioral: Physician management

INTERVENTIONS:
Behavioral: Early Direct Access Physical Therapy — Physical Therapy management including Manual therapy, Exercise, and education including cognitive behavioral therapy.
  Other Names: Physiotherapy management
  Arms: Early Direct Access Physical Therapy
Behavioral: Physician management — Physician management including advice, medication, and referral to physical therapy or other provider.
  Arms: Physician management

SUMMARY:
The purpose of this study is to determine whether seeing a physical therapist first compared with seeing a physician first is more clinically and cost effective in an occupational setting for acute musculoskeletal conditions.

DETAILED DESCRIPTION:
Traditionally, when individuals sustain a musculoskeletal injury and require physical therapy intervention, a referral is obtained from a physician to prescribe therapy. Currently, for non-work related injuries, 48 out of the 50 United States are "direct access physical therapy states" meaning a consumer can be evaluated and treated by a physical therapist directly without physician referral. The number of direct access states is much less for work-related injuries, with only 17 of the 50 United States practice acts permitting direct access, and of these, most insurance companies still require a physician referral for reimbursement. A previous systematic review of the literature on this topic suggests that requiring a referral is associated with more drug prescriptions, more imaging ordered, and higher costs to the patient and health care system with no advantage in health outcomes. However, the cited studies were of low quality (i.e. below Level 1 evidence), so a high quality study with strict experimental controls is still necessary.

This project proposes to conduct a blinded randomized controlled trial to determine if a "direct access physical therapy portal of entry" is more effective than a "physician portal of entry" in decreasing total episode cost and improving outcomes for individuals with a recent onset of musculoskeletal conditions. The project's definition of musculoskeletal pain is any "mechanical" spine or extremity pain from either a work condition (workers compensation) or a non-work related condition. The project investigators plan to recruit potential subjects directly from Temple University employees and supervisors. Subjects who consent to and pass a baseline screening will be randomized to one of two groups: direct access physical therapy management or Employee Health physician management. All PT and physician providers will be "study providers". Subjects randomized to direct access physical therapy will be evaluated and treated by a physical therapist. If the presentation requires further work up, the therapist will refer the patient for imaging or specialty consult. Subjects randomized to the Employee Health physician will receive a similar evaluation ordering relevant work up, and if appropriate, the physician will refer the patient to a physical therapist. Health outcomes for the two groups will be compared with a mixed-model repeated measures analysis at 1 month after enrollment. Total episode cost and medical utilization will be compared at one year after enrollment.

If this direct access "Temple University model" is feasible and effective for managing compensated and non-compensated musculoskeletal conditions, it could serve as a paradigm for other universities to implement across the United States. Furthermore, this study would be the first data set in the literature that studied a physical therapy direct access model for evaluation and treatment of employees with "workers-compensation" conditions in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Temple University Employees who speak English sufficiently to understand informed consent.
* Has a primary complaint that is potentially of neuro-musculoskeletal origin. This is defined by a primary complaint of pain, numbness, or decreased function due to symptoms within regions of spine, shoulder, elbow, wrist/hand pain, pelvic/SI, hip, knee, or ankle pain, temporomandibular joint pain, or headaches. The complaint could be work related (workers compensation) or non-work related. This definition does not include abrasions, contusions, etc. that result in pain but do not affect the employee's function.
* Age greater than or equal to 18 years old.
* Employee's primary complaint began ≤3 months upon initial study screening. This could include a recent exacerbation (within ≤3 months onset) of a condition with a history of previous episodes. If the patient reports more than one complaint, all complaints will be addressed in the study with intervention that began within the ≤3 month timeframe.

Exclusion Criteria:

* Met with another medical provider for advice for the condition prior to study enrollment (including physical therapist, chiropractor, physician, surgeon, physician-assistant, or nurse, etc.).
* Medical history of surgery for a prior episode of complaint.
* Any major psychiatric disease in their past medical history.
* Red flags cannot be ruled out during the medical screening examination (e.g., cauda equina compression, inflammatory arthritis, malignancy, fracture, serious illness or comorbidity). Any musculoskeletal injuries that can be managed by a physical therapist will not be excluded (radiculopathy, potential ACL tear, peripheral nerve entrapments, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2018-04-28 (Estimated); Study Completion 2018-04-28 (Estimated)

PRIMARY OUTCOMES:
Total Episode Cost and codes billed affecting cost | 1 year post study enrollment
  Reimbursed amounts related to initial presenting condition of interest including physical therapy, diagnostics, and all medical interventions (Medication prescriptions, physical therapy visits, physician office visits, specialty visits, imaging ordered, injections performed, number of surgeries performed)

SECONDARY OUTCOMES:
PROMIS, 10 item-Physical Function Questionnaire | 1 month post enrollement
  Self report questionnaire to assess function, quality of life
Patient-Specific Functional Scale (PSFS) | 1 month post enrollment
  Self report questionnaire (not region specific)
Pain Catastrophizing Score (PCS) | 1 month post enrollment
  Self-report standardized questionnaire, Theorized mediator
Pain Self-efficacy questionnaire (PSEQ) | 1 month post enrollment
  Self-report standardized questionnaire, Theorized mediator
Patient Satisfaction | 1 month post enrollment
  Self report rating from 0-10
Patient Acceptable Symptom State (PASS) | 1 month post enrollment
  Yes or No response to a written question if their current state is acceptable to patient.
Harm | 1 month post enrollment
  complaints voiced to the Workers Compensation Director, adverse events reported in the chart (defined as an undesirable result of the PT evaluation, diagnosis, or prescribed intervention resulting in any short-term or permanent morbidity unexpected for patients with a like clinical presentation), and litigation claims filed.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi A Ojha, DPT, Principal Investigator — Temple University
Locations (1):
- Temple University Employee Health, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fritz JM, Childs JD, Wainner RS, Flynn TW. Primary care referral of patients with low back pain to physical therapy: impact on future health care utilization and costs. Spine (Phila Pa 1976). 2012 Dec 1;37(25):2114-21. doi: 10.1097/BRS.0b013e31825d32f5. PMID 22614792
- [Result] Ojha HA, Snyder RS, Davenport TE. Direct access compared with referred physical therapy episodes of care: a systematic review. Phys Ther. 2014 Jan;94(1):14-30. doi: 10.2522/ptj.20130096. Epub 2013 Sep 12. PMID 24029295
- [Result] Wand BM, Bird C, McAuley JH, Dore CJ, MacDowell M, De Souza LH. Early intervention for the management of acute low back pain: a single-blind randomized controlled trial of biopsychosocial education, manual therapy, and exercise. Spine (Phila Pa 1976). 2004 Nov 1;29(21):2350-6. doi: 10.1097/01.brs.0000143619.34308.b4. PMID 15507794
- [Result] Zigenfus GC, Yin J, Giang GM, Fogarty WT. Effectiveness of early physical therapy in the treatment of acute low back musculoskeletal disorders. J Occup Environ Med. 2000 Jan;42(1):35-9. doi: 10.1097/00043764-200001000-00010. PMID 10652686
- [Derived] Ojha HA, Fritz JM, Malitsky AL, Wu J, Weiner MG, Brandi JA, Rhon DI, Mobo BHP, Fleming KM, Beidleman RR, Wright WG. Comparison of Physical Therapy and Physician Pathways for Employees with Recent Onset Musculoskeletal Pain: A Randomized Controlled Trial. PM R. 2020 Nov;12(11):1071-1080. doi: 10.1002/pmrj.12382. Epub 2020 May 23. PMID 32281269
- See also: Direct Access PT model in Nova Scotia for occupational soft tissue injuries — http://www.directaccesssummit.com/studies/1.pdf